CLINICAL TRIAL: NCT00542282
Title: Evaluation of Vibration Response Imaging (VRI) in Chronic Obstructive Pulmonary Disease and Asthma Patients Before and After Bronchodilators
Brief Title: Vibration Response Imaging in Chronic Obstructive Pulmonary Disease and Asthma
Status: Completed | Type: Observational
Sponsor: Deep Breeze (Industry)
Responsible Party: Merav Gat/VP Clinical Affairs, Deep Breeze
Other Study IDs: DB033
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Last update posted 2009-06-16 (Estimated); Status verified 2009-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; Asthma
Keywords: lung sounds,; airway obstruction,; asthma,; auscultation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Respiratory Sounds; Airway Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1, 2, 3: known moderate to severe COPD, known moderate or severe Asthma, suspected obstructive moderate to severe airways disease

SUMMARY:
Obstructive lung disease is usually a differential diagnostic consideration when a patient presents with breathlessness or cough. Spirometry is the key diagnostic test used to confirm airflow obstruction particularly in the primary care setting. Airflow obstruction that completely resolves after administration of a bronchodilator, by definition, excludes a diagnosis of COPD. Evaluation of obstructive lung disease must include pulmonary function testing; bronchoreversibility testing is an adjunct in differentiating between asthma and COPD. Bronchoreversibility cannot serve as an absolute diagnostic criterion for separating asthma from COPD.

Vibration response imaging (VRI) technology provides a simple, radiation-free method to image the lungs, by visualizing vibration energy (lung sounds) emitted during respiration cycle. In this study, regional quantitative and qualitative information on vibration response is compared with spirometry in assessing lungs function of COPD and Asthma patients.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to read, understand, and provide written Informed Consent
* Male or Female in the age range of 18-85 years
* Patients referred for evaluation of known or suspected obstructive airways disease.
* Subject is referred for pulmonary function testing with pre-and post- bronchodilator
* BMI > 21
* Patients who are treated with Bronchodilators should go through a washout period prior the VRI procedure according to the Pulmonary Function Laboratory protocol.
* Stable clinical condition at study baseline evaluation.

Exclusion Criteria:

* Chest wall deformation
* Spine deformation (including severe scoliosis)
* Hirsutism
* Potentially contagious skin lesion on the back
* Skin lesion that would interfere with sensor placement
* Pregnant or lactating females.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are either suspected of pulmonary obstruction or already diagnosed and are scheduled to perform a spirometry test with pre and post administration of bronchodilators will be enrolled in this study
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2006-11; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The primary study objective is evaluation of the VRI qualitative and quantitative assessment before and after spirometry with bronchodilators. | One day

SECONDARY OUTCOMES:
The secondary objective is correlating the VRI evaluations with lung function test results | One day

CONTACTS AND LOCATIONS:
Overall Officials: Kalpalatha K Guntupalli, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Background] van Schayck CP, Chavannes NH. Detection of asthma and chronic obstructive pulmonary disease in primary care. Eur Respir J Suppl. 2003 Jan;39:16s-22s. doi: 10.1183/09031936.03.00040403. PMID 12572697
- [Background] Dellinger RP, Parrillo JE, Kushnir A, Rossi M, Kushnir I. Dynamic visualization of lung sounds with a vibration response device: a case series. Respiration. 2008;75(1):60-72. doi: 10.1159/000103558. Epub 2007 Jun 4. PMID 17551264
- [Background] Dellinger RP, Jean S, Cinel I, Tay C, Rajanala S, Glickman YA, Parrillo JE. Regional distribution of acoustic-based lung vibration as a function of mechanical ventilation mode. Crit Care. 2007;11(1):R26. doi: 10.1186/cc5706. PMID 17316449